CLINICAL TRIAL: NCT01232179
Title: Comparison Between Result and Side Effects of Treatment of Prolifrative Diabetic Retinopaty by Conventional and Extended Targeted Pan Retinal Photocoagolation
Brief Title: Comparison of Two Laser Therapy Methods for PDR
Acronym: PDR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Masoud Soheilian, Ophthalmic Research center
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 88100
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-10

CONDITIONS: Proiriftrative Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- conventional prp (Active Comparator)
  Interventions: Procedure: conventional prp
- targeted PRP (Active Comparator)
  Interventions: Procedure: targeted prp

INTERVENTIONS:
Procedure: conventional prp — pan retinal photocoagulation
  Arms: conventional prp
Procedure: targeted prp — 1200-1600 spot in far periphery retin, anterior equator
  Arms: targeted PRP

SUMMARY:
Proliferative diabetic retinopathy (PDR) is treated with conventional pan retinal photocoagulation (PRP) which can improve the visual prognosis in this complication significantly. However , the treatment may also resulting adverse effects such as blurring of central vision, visual field constriction and disturbance in dark adaptation and contrast vision. Extended targeted retinal coagulation (TRP) to the ischemic areas may cause regression of the neovascularization while minimizing some of the risks and complication associated of treatment of PDR with these two methods.

ELIGIBILITY:
Inclusion Criteria:

* patients with PDR condidate for photocoagulation teraphy
* Pupil with dilatasion≥6mm
* without privious treatment with anti VEGF drugs 3months before study
* without privious vitroretinal sugery
* without privoius lasertraphy

Exclusion Criteria:

* To have NVI cricteria with increase of inraocular pressure
* to have cataract or vitrus leakage which prevent lasertraphy
* pupil smaller that 6mm
* traditional retinal detachment
* privious treatment with anti VEGF drugs 3months before study
* privious PRP
* patient unable to get wide field FAG

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2010-10; Primary Completion 2011-04 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
no leakage in widefield fluorescin angiography | 3 months after lasertraphy

CONTACTS AND LOCATIONS:
Locations (1):
- Labbafinejad medical center, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Nikkhah H, Ghazi H, Razzaghi MR, Karimi S, Ramezani A, Soheilian M. Extended targeted retinal photocoagulation versus conventional pan-retinal photocoagulation for proliferative diabetic retinopathy in a randomized clinical trial. Int Ophthalmol. 2018 Feb;38(1):313-321. doi: 10.1007/s10792-017-0469-7. Epub 2017 Feb 6. PMID 28168567